CLINICAL TRIAL: NCT01447628
Title: What is the Effect of Intravenous Iron Supplementation on Cardiopulmonary Haemodynamics, Exercise Capacity and Quality of Life in Patients With IPAH and Iron Deficiency?
Brief Title: IV Iron Replacement for Iron Deficiency in Idiopathic Pulmonary Arterial Hypertension (IPAH) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO1811
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Arterial Hypertension; Iron Deficiency
Keywords: Idiopathic pulmonary arterial hypertension (IPAH); Iron deficiency
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Iron Deficiencies; Familial Primary Pulmonary Hypertension | interventions — Sodium Chloride; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferinject or CosmoFer followed by Placebo (Active Comparator): IV iron formulation used in Europe - Ferinject - given over 15 minutes
  IV iron formulation used in China - CosmoFer - over a period of 4 to 6 hours
  IV Iron given at Week 0, Placebo (saline) given at Week 12.
  Interventions: Drug: Saline; Drug: Ferinject or CosmoFer
- Placebo followed by Ferinject or CosmoFer (Placebo Comparator): Placebo comparator
  Placebo (saline) given at Week 0, IV Iron given at Week 12.
  Interventions: Drug: Saline; Drug: Ferinject or CosmoFer

INTERVENTIONS:
Drug: Saline — intravenous, no active drug
  Other Names: Placebo
Drug: Ferinject or CosmoFer — Intravenous, 1000 mg iron
  Other Names: Intravenous Iron

SUMMARY:
This study will establish whether intravenous iron replacement has clinical benefit in idiopathic pulmonary arterial hypertension.

A 24-week double-blind, randomised, placebo-controlled, crossover study will investigate whether a single dose of 1g of Ferinject® or CosmoFer improves cardiopulmonary haemodynamics, exercise capacity and quality of life and is well-tolerated.

IV iron formulation used in Europe - Ferinject IV iron formulation used in China - CosmoFer

DETAILED DESCRIPTION:
These results represent the outcome of two separate clinical trials which were conducted in collaboration, led by Imperial College and Fuwai, China respectively. The protocols were analogous, although in China Endurance Cardio-Pulmonary Exercise Testing (CPET) was not done and instead of Ferinject/Placebo being infused over 15 minutes, Cosmofer/Placebo was infused over 4-6 hours.

The study analyses were performed as Intention to Treat, except for patients 6009-6017 as described below. The study was a cross-over design and results are presented for 2 groups based on the participants' study timepoint, and presented separately for the two study datasets (Europe and Fuwai). A meta-analysis was conducted for the combined data where possible and the relevant p-values have been provided.

Iron results in the European dataset are taken from blood results which were collected centrally and analysed by one laboratory at Imperial College London. N-Terminal B-type natriuretic peptide (NT-PRO-BNP) and Soluble Transferrin Receptors (STFR) were not done at Fuwai.

The study was conducted according to Good Clinical Practice (GCP), but there were some missing data (imputed using multiple imputation techniques), and also some significant protocol deviations which are summarised below.

Six participants (2003, 3004, 4002-4005) had their endurance CPETs set at incorrect workloads which differed significantly from that achieved at the baseline incremental CPET. These data were therefore treated as missing, and relevant values imputed as per the statistical analysis plan.

Visit 5 CPETs for participants 1008 (Incremental CPET 12 weeks later) 1018 (Endurance CPET 13 days later) and 1019 (Incremental CPET 15 days later) were performed outside the protocol-specified window.

Participant 1014 received placebo at both treatment visits in error. Participant 6017 suffered a suspected allergic reaction to their first infusion and was withdrawn from the study. There was a systemic error where participants 6009-6016 received the opposite to their random-assigned treatment at each time point. These participants were analysed according to the treatment actually received, rather than that originally assigned by randomisation.

ELIGIBILITY:
* Males or females aged between 16-75 years old
* Pulmonary Arterial Hypertension (PAH) which is idiopathic, heritable or associated with anorexigens.
* Iron deficiency (TfR levels > 28.1 nmol/l, where sTfR analysis is available, Ferritin < 37 ug/l; transferrin saturations < 16.4%; iron < 10.3 umol/l)
* Documented diagnosis of PAH by right heart catheterisation performed at any time prior to Screening showing: resting mean pulmonary artery pressure >25mmHg, pulmonary capillary wedge pressure =/< 15 mm Hg and normal or reduced cardiac output;
* 6 minute walking distance greater than 50m at entry;
* Stable on an unchanged PAH therapeutic regime (any combination of endothelin receptor antagonist, phosphodiesterase inhibitor or prostacyclin analogue) for at least 1 month.
* Able to provide written informed consent prior to any study-mandated procedures
* Female subjects of child-bearing potential are eligible to participate if they agree to use one of the following contraception methods:
* Abstinence
* Contraceptive methods with a failure rate of < 1%:
* Oral contraceptive, either combined or progestogen alone;
* Injectable progestogen;
* Implants of levonorgestrel;
* Estrogenic vaginal ring;
* Percutaneous contraceptive patches;
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the <1% failure rate as stated in the product label;
* Male partner(s) sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study;
* Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus vaginal spermicidal agent (foam/gel/film/cream/suppository).

Exclusion criteria

* Unable to provide informed consent.
* Clinically-significant renal disease (Creatinine clearance < 30 ml/min per 1.73 m2 calculated from Chronic Kidney Disease-Epidemiology Collaboration (CKD-Epi) http://www.qxmed.com/renal/Calculate-CKD-EPI-GFR.php) or liver disease (including serum transaminases > 3 times upper limit of normal).
* Haemoglobin concentration <10 g/dl.
* Patients will be excluded if any single parameter (iron, ferritin or transferrin saturation) exceeds 1x upper limit of normal (ULN) in the local lab reference range.
* Patients with moderate to severe hypophosphatemia as defined as <0.65mmol/L
* Known to have haemoglobinopathy e.g. sickle cell disease, thalassaemia.
* Admission to hospital related to PAH or change in PAH therapy within 1 month prior to Screening.
* Evidence of left ventricular disease or significant lung disease on high-resolution Computed Tomography (CT) scanning or lung function as judged by the investigator
* Acute or chronic infection or inflammation.
* Significant uncontrolled asthma as judged by the investigator, eczema or atopic allergies.
* Females who are lactating or pregnant.
* Individuals known to have Human Immunodeficiency Virus (HIV), Hepatitis B or C or Creutzfeld-Jakob disease.
* Known hypersensitivity to Ferinject® or any of its excipients.
* Evidence of disturbances in utilisation of iron.
* Significant blood loss (e.g. Gastro-intestinal bleed) within the last 3 months or history of menorrhagia.
* Unable to perform a Cardiopulmonary Exercise Test i.e. due to syncope or musculoskeletal factors.
* Patients who have received an investigational medicinal product within 30 days of entering the baseline visit

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke Howard, DPhil, FRCP, Principal Investigator — Imperial College London
Locations (5):
- Fuwai Hospital, Beijing, China
- Justus-Liebig University, Giessen, Germany
- United Kingdom (3):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Hammersmith Hospital, Imperial College NHS Trust, London
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howard LSGE, He J, Watson GMJ, Huang L, Wharton J, Luo Q, Kiely DG, Condliffe R, Pepke-Zaba J, Morrell NW, Sheares KK, Ulrich A, Quan R, Zhao Z, Jing X, An C, Liu Z, Xiong C, Robbins PA, Dawes T, de Marvao A, Rhodes CJ, Richter MJ, Gall H, Ghofrani HA, Zhao L, Huson L, Wilkins MR. Supplementation with Iron in Pulmonary Arterial Hypertension. Two Randomized Crossover Trials. Ann Am Thorac Soc. 2021 Jun;18(6):981-988. doi: 10.1513/AnnalsATS.202009-1131OC. PMID 33735594

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The groups are separated into Europe and China, because a different Investigational Medicinal Product (IMP) was used and outcome measures were analysed separately.
Groups:
- Ferinject Followed by Placebo (Europe): IV iron formulation used in Europe - Ferinject (Intravenous, 1000 mg iron)- given over 15 minutes followed by Placebo given as 1000mg saline according to randomisation.
  Ferinject administered at week 0, placebo (saline) administered at week 12.
- Placebo Followed by Ferinject (Europe): IV iron formulation used in Europe - Ferinject (Intravenous, 1000 mg iron)- given over 15 minutes or Placebo given as 1000mg saline according to randomisation.
  Placebo (saline) administered at week 0, Ferinject administered at week 12.
- Cosmofer Followed by Placebo (China): IV iron formulation used in China was CosmoFer - given intravenously over a period of 4 to 6 hours
  Cosmofer administered at week 0, placebo (saline) administered at week 12.
- Placebo Followed by Cosmofer (China): IV iron formulation used in China was CosmoFer - given intravenously over a period of 4 to 6 hours
  Placebo (saline) administered at week 0, Cosmofer administered at week 12.
Period: Week 0 to Week 12 (1st Intervention)
Arm/Group | Ferinject Followed by Placebo (Europe) | Placebo Followed by Ferinject (Europe) | Cosmofer Followed by Placebo (China) | Placebo Followed by Cosmofer (China)
Started | 19 | 20 | 12 (Randomisation error meant the arms were not balanced- refer to protocol description for full details) | 5 (Randomisation error meant the arms were not balanced- refer to protocol description for full details)
Completed | 19 | 20 | 12 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Week 12 to Week 24 (2nd Intervention)
Arm/Group | Ferinject Followed by Placebo (Europe) | Placebo Followed by Ferinject (Europe) | Cosmofer Followed by Placebo (China) | Placebo Followed by Cosmofer (China)
Started | 19 | 20 | 12 | 4
Completed | 19 | 20 | 12 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was conducted as a cross-over study, but for the statistical analysis, data for participants were grouped by timepoint to provide an overall comparison between active and placebo treatment. Hence each analysis group contains all participants, as all received both IMP and placebo.
Groups:
- European Dataset: IV iron (1000 mg) formulation used in Europe - Ferinject - given over 15 minutes
  Saline: intravenous, no active drug
- China Dataset: IV iron (1000mg) formulation used in China - CosmoFer - over a period of 4 to 6 hours
  Saline: intravenous, no active drug
- Total: Total of all reporting groups
Arm/Group | European Dataset | China Dataset | Total
Number analyzed (Participants) | 39 | 17 | 56
Age, Continuous [Mean (Full Range); unit: years] | 49.4 [18 to 75] | 32.58 [18 to 54] | 44.3 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 15 | 44
  Male | 10 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 17 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 0 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 0 | 17 | 17
  United Kingdom | 34 | 0 | 34
  Germany | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity - Endurance
Description: Time measured in seconds from start to end of the endurance bicycle cardiopulmonary exercise testing at 80% of the peak work rate. Peak work rate is determined by that achieved at the baseline incremental cardiopulmonary exercise test (CPET).
  Note that this was the primary end-point of the European study. Endurance CPET was not done in China.
Time Frame: 12 Weeks post study treatment
Population: Intention to treat (ITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Groups:
- Ferinject Group (Europe): IV iron formulation used in Europe - Ferinject (Intravenous, 1000 mg iron)- given over 15 minutes
  This group provides the outcome measurements for participants following their infusion of Ferinject whether this was at the first or second timepoint
- Placebo Group (Europe): Placebo (saline) given intravenously over 15 minutes.
  This group provides the outcome measurements for participants following their infusion of Placebo whether at the first or second timepoint
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
Seconds | 315.44 [274.68 to 356.20] | 302.89 [260.09 to 345.69]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.6039, Mixed Models Analysis

2. Primary Outcome: Change in Resting Pulmonary Vascular Resistance (PVR)
Description: To be measured by cardiac catheterisation in wood units.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: Wood units
Groups:
- Ferinject Group (Europe): IV iron formulation used in Europe - Ferinject (Intravenous, 1000 mg iron)- given over 15 minutes
  This group provides the outcome measurements for participants following their infusion of Ferinject, whether this was at the first or second timepoint
- Placebo Group (Europe): Placebo (saline) given intravenously over 15 minutes.
  This group provides the outcome measurements for participants following their infusion of Placebo, whether this was at the first or second timepoint
- Cosmofer Group (China): This group provides the outcome measurements for participants following their infusion of CosmoFer, whether this was at the first or second timepoint.
  IV iron formulation used in China was CosmoFer - given intravenously over a period of 4 to 6 hours
- Placebo Group (China): This group provides the outcome measurements for participants from the Fuwai site following their infusion of Placebo (saline, infused over 4-6hrs), whether this was at the first or second timepoint.
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
Wood units | 7.69 [5.71 to 9.17] | 5.15 [3.61 to 7.27] | 11.70 [9.16 to 14.04] | 9.5 [6.25 to 13.81]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.0747, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.7990, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); This is a combination of the p-values from the separate analyses of each data set; Test type: Superiority; p = 0.2111, Mixed Models Analysis

3. Secondary Outcome: Oxygen Consumption (VO2) Level at Peak 12 Weeks After Study Treatment
Description: Level of VO2 at peak measured during incremental cardio-pulmonary exercise testing
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: Litres per minute
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
Litres per minute | 1.17 [1.10 to 1.22] | 1.13 [1.08 to 1.21] | 0.93 [0.87 to 1.00] | 0.94 [0.84 to 0.97]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.6583, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9166, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.6631, Mixed Models Analysis

4. Secondary Outcome: Oxygen Consumption (VO2) at Metabolic Threshold
Description: Level of VO2 at metabolic threshold measured during incremental cardio-pulmonary exercise test
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: Litres per minute
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
Litres per minute | 0.78 [0.73 to 0.82] | 0.77 [0.73 to 0.82] | 0.66 [0.58 to 0.76] | 0.69 [0.59 to 0.77]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.4039, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9144, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9959, Mixed Models Analysis

5. Secondary Outcome: Ventilation / Volume of Exhaled Carbon Dioxide (VE/VCO2 Slope)
Description: VE/VCO2 slope measured during incremental cardio-pulmonary exercise testing
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: l/min/l/min
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
l/min/l/min | 41.15 [39.43 to 42.93] | 42.35 [40.58 to 44.07] | 35.06 [30.66 to 39.31] | 36.27 [31.21 to 39.78]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.1788, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.7795, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.414, Mixed Models Analysis

6. Secondary Outcome: Oxygen Consumption (VO2) / Work Rate (WR) Slope
Description: Level of VO2 / WR Slope measured during incremental cardio-pulmonary exercise testing
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: ml/min/watt
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
ml/min/watt | 8.12 [7.50 to 8.71] | 8.04 [7.46 to 8.68] | 5.97 [5.15 to 6.77] | 6.04 [5.15 to 6.77]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.8688, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9999, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.991, Mixed Models Analysis

7. Secondary Outcome: Peak Oxygen (O2) Pulse Rate
Description: O2 pulse rate (amount of oxygen consumed per heart beat) at peak measured during incremental cardio-pulmonary exercise test
Time Frame: 12 weeks post study treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/beat
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
ml/beat | 13.30 [10.00 to 16.59] | 11.92 [8.30 to 15.54] | 6.55 [6.02 to 7.01] | 6.36 [5.79 to 6.79]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.5465, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.4298, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.5451, Mixed Models Analysis

8. Secondary Outcome: Oxygen Consumption (VO2) at the End of Endurance Cardio-pulmonary Exercise Test (CPET)
Description: Level of VO2 measured at end of endurance cardio-pulmonary exercise test. Note that endurance CPET was not done in China, so this is reported only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres per minute
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
Litres per minute | 4.25 [3.50 to 5.01] | 4.49 [3.71 to 5.28]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Note that Endurance CPET was not done in China, hence only European data provided; Test type: Superiority; p = 0.6241, Mixed Models Analysis

9. Secondary Outcome: Oxygen Consumption (VO2) at 3 Minutes
Description: Level of VO2 measured at 3 minutes into endurance cardio-pulmonary exercise test (CPET) Note that endurance CPET was not done in China, hence results are presented only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres per minute
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
Litres per minute | 1.29 [0.98 to 1.60] | 1.14 [0.81 to 1.48]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.4758, Mixed Models Analysis

10. Secondary Outcome: Iron Indices: Serum Iron
Description: Measurement of serum iron
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
umol/L | 17.15 [15.42 to 18.64] | 15.48 [13.94 to 17.17] | 15.81 [12.29 to 19.25] | 14.31 [9.83 to 16.79]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.2050, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.1993, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.1993, Mixed Models Analysis

11. Secondary Outcome: Iron Indices: Transferrin Saturations
Description: Measurement of serum transferrin saturations. The saturation measures the iron concentration as a proportion of the iron binding capacity of transferrin.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: percentage of iron occupied transferrin
Groups:
- Ferinject European Dataset: Active IMP: Measure of transferrin saturations in European patients receiving active treatment.
- Ferinject European Dataset: Placebo Arm: Measure of transferrin saturations at 12 weeks in European patients receiving placebo
- Cosmofer: China Dataset Active: Measure of transferrin saturations in China patients receiving Cosmofer
- Placebo: China Dataset: Measure of transferrin saturations in China patients receiving Placebo
Arm/Group | Ferinject European Dataset: Active IMP | Ferinject European Dataset: Placebo Arm | Cosmofer: China Dataset Active | Placebo: China Dataset
Number analyzed (Participants) | 39 | 39 | 17 | 17
percentage of iron occupied transferrin | 26.2 [22.96 to 28.89] | 22 [19.21 to 25.12] | 26.81 [20.81 to 31.51] | 22.88 [15.27 to 26.00]
Statistical Analysis 1: Comparison: Ferinject European Dataset: Active IMP vs Ferinject European Dataset: Placebo Arm; Test type: Superiority; p = 0.0610, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer: China Dataset Active vs Placebo: China Dataset; Test type: Superiority; p = 0.0641, Mixed Models Analysis

12. Secondary Outcome: Iron Indices: Ferritin
Description: Measured level of serum ferritin
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: ug/L
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
ug/L | 150.32 [118.63 to 175.51] | 92.74 [66.08 to 122.88] | 135.06 [122.79 to 165.29] | 65.5 [44.27 to 86.77]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.0003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p < 0.0001, Mixed Models Analysis

13. Secondary Outcome: Iron Indices: Soluble Transferrin Receptors (sTfR)
Description: Measure of serum sTfR level. Note that this was not measured in China, hence is reported only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
nmol/L | 28.37 [25.73 to 31.72] | 37.25 [34.02 to 40.00]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p < 0.0001, Mixed Models Analysis

14. Secondary Outcome: 6 Minute Walk Test: Distance Walked
Description: Distance in metres walked during standardised and validated 6 minute walk test
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: Metres
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
Metres | 426.03 [411.57 to 440.20] | 424.3 [410.06 to 438.70] | 478 [448.96 to 523.59] | 474.19 [443.73 to 518.37]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.8093, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.6300, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.8533, Mixed Models Analysis

15. Secondary Outcome: 6 Minute Walk Test: Borg Dyspnoea Score After Test
Description: Participant reported score on the modified Borg Dyspnoea scale (0-10) following 6 minute walk test. Higher scores indicate worsened dyspnoea.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
units on a scale | 3.24 [2.75 to 3.75] | 3.68 [3.18 to 4.17] | 1.38 [0.72 to 2.00] | 1.28 [0.66 to 1.93]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.0725, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.8572, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.2348, Mixed Models Analysis

16. Secondary Outcome: Iron Indices: N-terminal Pro B-type Natriuretic Peptide (NT-pro-BNP)
Description: Measured level of NT-pro-BNP in blood sample. Note that this was not measured in China, hence is presented only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: fmol/ml
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
fmol/ml | 307.64 [186.47 to 437.62] | 394.94 [297.52 to 548.39]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.1115, Mixed Models Analysis

17. Secondary Outcome: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR Questionnaire): Symptom Score
Description: Participant self reported symptom score using the CAMPHOR questionnaire (0-25). Scores for symptoms range from 0-25, with higher scores indicating worse symptoms.
  Note that this was not measured in China, hence is presented only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
score on a scale | 7.94 [6.99 to 8.89] | 7.94 [7.02 to 8.89]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.9790, Mixed Models Analysis

18. Secondary Outcome: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR Questionnaire): Activity Score
Description: Participants' self reported score of their own level of activity based on the CAMPHOR questionnaire.
  Activity scores range from 0-30, with higher scores indicating more physical limitations Note that this was not measured in China, hence is presented only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
units on a scale | 9.12 [8.14 to 10.07] | 9.18 [8.25 to 10.16]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.7702, Mixed Models Analysis

19. Secondary Outcome: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR Questionnaire): QoL Score
Description: Quality of Life score based on the Cambridge Pulmonary Hypertension Outcomes Review (CAMPHOR) questionnaire (0-25).
  Scores for QoL range from 0-25, with higher scores indicating worse quality of life Note that this was not measured in China, hence is presented only for the European dataset.
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe)
Number analyzed (Participants) | 39 | 39
units on a scale | 7.58 [6.38 to 8.69] | 7 [5.91 to 8.16]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.2219, Mixed Models Analysis

20. Secondary Outcome: Mean Right Atrial Pressure (Cardiac Catheter)
Description: Mean right atrial pressure at rest measured by cardiac catheter
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
mmHg | 6.56 [5.40 to 9.23] | 10.12 [7.17 to 11.21] | 6.67 [4.55 to 7.91] | 4.5 [3.21 to 8.48]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.1777, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.7889, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.4156, Mixed Models Analysis

21. Secondary Outcome: Oxygen Consumption (VO2) Level at Peak
Description: VO2 at peak of Incremental Cardio-pulmonary exercise test in ml/min/kg
Time Frame: 12 weeks post study treatment
Measure: Mean (95% Confidence Interval); unit: ml/min/kg
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
ml/min/kg | 15.10 [14.10 to 15.58] | 14.67 [14.20 to 15.68] | 14.53 [12.83 to 16.68] | 14.36 [11.21 to 15.09]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.7625, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.2262, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.4756, Mixed Models Analysis

22. Secondary Outcome: Oxygen Consumption (VO2) at Metabolic Threshold
Description: VO2 at Metabolic Threshold measured during incremental cardio-pulmonary exercise test
Time Frame: 12 weeks post treatment
Measure: Mean (95% Confidence Interval); unit: ml/min/kg
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
ml/min/kg | 10.01 [9.45 to 10.46] | 9.99 [9.52 to 10.53] | 10.91 [9.98 to 12.06] | 11.2 [9.77 to 11.86]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.7711, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.7806, Mixed Models Analysis
Statistical Analysis 3: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9074, Mixed Models Analysis

23. Secondary Outcome: Stroke Volume (Cardiac Catheter)
Description: Measurement of stroke volume at rest by cardiac catheter at 12 weeks post treatment
Time Frame: 12 weeks post treatment
Measure: Mean (95% Confidence Interval); unit: mililitres
Arm/Group | Ferinject Group (Europe) | Placebo Group (Europe) | Cosmofer Group (China) | Placebo Group (China)
Number analyzed (Participants) | 39 | 39 | 17 | 17
mililitres | 77.87 [77.41 to 102.05] | 99.71 [75.86 to 102.02] | 55.11 [49.57 to 61.15] | 54.65 [45.22 to 63.17]
Statistical Analysis 1: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe) vs Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.9504, Mixed Models Analysis
Statistical Analysis 2: Comparison: Ferinject Group (Europe) vs Placebo Group (Europe); Test type: Superiority; p = 0.8666, Mixed Models Analysis
Statistical Analysis 3: Comparison: Cosmofer Group (China) vs Placebo Group (China); Test type: Superiority; p = 0.8104, Mixed Models Analysis

24. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Right Ventricular End-diastolic Volume
Description: Cardiac MRI: Right ventricular end-diastolic volumes
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: mililitres
Groups:
- Cardiac MR Dataset: Active Treatment: This group includes all participants in the Europe and China Dataset that volunteered to the optional cardiac MR that received active treatment
- Cardiac MR Dataset: Placebo: This group includes all participants in the Europe and China Dataset that volunteered to the optional cardiac MR that received Placebo
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
mililitres | 201.35 [195.26 to 207.44] | 203.06 [196.97 to 209.15]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.4478, Mixed Models Analysis

25. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Right Ventricular End Systolic Volume (RVESV)
Description: Cardiac MR: Right ventricular end systolic volume
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: mililitres
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
mililitres | 124.99 [120 to 129.98] | 126.31 [121.32 to 131.29]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.4590, Mixed Models Analysis

26. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Right Ventricular Stroke Volume (RVSV)
Description: Right ventricular stroke volumes assessed by cardiac MRI scan
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: mililitres
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
mililitres | 76.46 [73.56 to 80.13] | 76.84 [73.56 to 80.13]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.8086, Mixed Models Analysis

27. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Right Ventricular Ejection Fraction (RVEF)
Description: Cardiac MR: Right ventricular ejection fractions
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
percentage | 39.89 [38.55 to 41.23] | 39.64 [38.31 to 40.98]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.6944, Mixed Models Analysis

28. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Left Ventricular End Diastolic Volume (LVEDV)
Description: Cardiac MR: Left Ventricular End Diastolic Volume
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Mililitres
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
Mililitres | 117.36 [113.47 to 121.26] | 118.33 [114.43 to 122.22]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.585, Mixed Models Analysis

29. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Left Ventricular End Systolic Volume (LVESV)
Description: Cardiac MR: Left Ventricular End Systolic Volume
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Mililitres
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
Mililitres | 43.90 [41.84 to 45.96] | 44.43 [42.37 to 46.49]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.4619, Mixed Models Analysis

30. Secondary Outcome: Cardiac Magnetic Resonance Imaging: Left Ventricular Stroke Volume (LVSV)
Description: Cardiac MR: Left Ventricular Stroke Volume
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Mililitres
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
Mililitres | 43.90 [41.84 to 45.96] | 73.96 [69.98 to 77.95]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.7721, Mixed Models Analysis

31. Secondary Outcome: Cardiac Magnetic Resonance Imaging (MRI): Left Ventricular Ejection Fraction (LVEF)
Description: Cardiac MR: Left Ventricular Ejection Fraction
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
Percentage | 63.10 [61.38 to 64.81] | 62.94 [61.22 to 64.65]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.8332, Mixed Models Analysis

32. Secondary Outcome: Cardiac Magnetic Resonance Imaging: Left Ventricular Mass
Description: Cardiac MR: Left Ventricular Mass
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Grams
Arm/Group | Cardiac MR Dataset: Active Treatment | Cardiac MR Dataset: Placebo
Number analyzed (Participants) | 30 | 30
Grams | 72.82 [70.82 to 74.82] | 73.53 [71.53 to 75.53]
Statistical Analysis 1: Comparison: Cardiac MR Dataset: Active Treatment vs Cardiac MR Dataset: Placebo; Test type: Superiority; p = 0.2651, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events collected from consent until the final follow-up visit at week 24.
Groups:
- European Dataset: Iron: IV iron formulation used in Europe - Ferinject - given over 15 minutes
  Ferinject or CosmoFer: Intravenous, 1000 mg iron
  Time scale is within 12 weeks from Ferinject administration
- European Dataset: Placebo; China Dataset: Placebo: Placebo was 1000mg saline: intravenous, no active drug
  Time scale is within 12 weeks from saline administration
- European Dataset: Outside Window; China Dataset: Outside Window: AEs reported before intervention or more than 12 weeks following both Iron and Placebo.
- China Dataset: Iron: IV iron formulation used in China - CosmoFer - over a period of 4 to 6 hours
  Ferinject or CosmoFer: Intravenous, 1000 mg iron
  Time scale is within 12 weeks from Ferinject administration
Arm/Group | European Dataset: Iron | European Dataset: Placebo | European Dataset: Outside Window | China Dataset: Iron | China Dataset: Placebo | China Dataset: Outside Window
All-Cause Mortality (participants affected / at risk) | 26/39 | 28/39 | 13/39 | 3/17 | 4/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 4/39 | 3/39 | 1/39 | 0/17 | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 22/39 | 21/39 | 11/39 | 3/17 | 4/17 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | European Dataset: Iron (N=39) | European Dataset: Placebo (N=39) | European Dataset: Outside Window (N=39) | China Dataset: Iron (N=17) | China Dataset: Placebo (N=17) | China Dataset: Outside Window (N=17)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Line infection from Groshong line (Presented with pyrexia 39.7 degrees C. patient hospitalised, treated with antibiotics and fully recovered)
Hypophosphatemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Required hospitalisation
Haemorrhagic Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient fell and cut their face and nose which bled heavily. Patient on Warfarin at the time. Hospitalised and given CT scan and stiches.
Disease Progression (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Para-spinal haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection: Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Believed to be allergic-type reaction to IMP / placebo infusion. Patient suffered a rash and itchiness after 10 minutes of starting infusion. Recovered after administration of anti-allergic medications.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | European Dataset: Iron (N=39) | European Dataset: Placebo (N=39) | European Dataset: Outside Window (N=39) | China Dataset: Iron (N=17) | China Dataset: Placebo (N=17) | China Dataset: Outside Window (N=17)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Flu like symptoms (General disorders) | 7 (9) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 5 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Investigations) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated NT-Pro BNP (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysguesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Refer to the detailed study description in the protocol section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publications should be agreed in advance by the sponsor via the Chief Investigator. Publications will be written by Chief investigator with contributions from collaborating investigators acknowledged appropriately (e.g. via authorship). Trial agreements between sponsor and participating site provide full details of publication restrictions and review timelines.

DOCUMENTS (2):
  • Study Protocol (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT01447628/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT01447628/SAP_002.pdf